CLINICAL TRIAL: NCT05277116
Title: The Electronic Medical Records and GEnomics (eMERGE) Network Genomic Risk Assessment
Acronym: eMERGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Josh Peterson, Professor of Biomedical Informatics and Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 211043
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Genetic Disease
Keywords: Genomic Risk; Genomic Medicine; GIRA; Genome Informed Risk Assessment; Risk Report
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: All participants will receive a genome informed risk assessment (GIRA) report. Participants designated as high risk based on their genomic risks will be compared to those without such risks for each condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants receiving a Genome Informed Risk Assessment (GIRA) (Experimental): All participants and their health care providers will receive a Genome Informed Risk Assessment (GIRA) report.
  Interventions: Other: Genome Informed Risk Assessment (GIRA) report

INTERVENTIONS:
Other: Genome Informed Risk Assessment (GIRA) report — A Genome Informed Risk Assessment (GIRA) report that combines genetic (monogenic risks and polygenic risk scores), family history, and clinical risk information from participants.

SUMMARY:
The eMERGE Network embraces the opportunity to use new methods in genomic medicine, information science, and research participant engagement to identify people at very high risk for specific diseases and recommend individualized approaches to prevention and care. The investigators will conduct a prospective study, with diverse and underserved participants, across ten eMERGE study sites to evaluate clinical implementation of a Genome Informed Risk Assessment (GIRA) tool that combines genetic, family history, and clinical risk information from participants.

DETAILED DESCRIPTION:
The purpose of the study is to determine if providing a Genome Informed Risk Assessment (GIRA) will impact clinical actions taken by providers and patients to manage disease risk and the propensity of participants to develop a disease reported in the GIRA. New tools in Genomic Medicine - polygenic risk scores, monogenic genetic screening tests, platforms to capture family history, and advanced electronic phenotyping - offer the prospect of early identification of people at especially high risk of common diseases. The investigators developed methods to generate integrated genomic risk assessments for ten conditions; a plan to engage, recruit, and retain ~25,000 subjects to receive these assessments; and methods to study outcomes in those designated high risk and those designated non-high risk. By enhancing understanding of new methods to create and deliver integrated genomic risk assessments, this project will enable prevention and early treatment of people at high risk for common diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-75
* Children 3 to < 18
* Able to read or understand English or Spanish
* Able to provide a healthcare provider or clinician to receive results
* Willing to accept GIRA report

Exclusion Criteria:

* Inability to provide consent
* Transplant (solid organ or bone marrow) or transfusion within 8 weeks
* Research staff and investigators in eMERGE
* Not a patient at parent institution

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26877 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of new health care actions after return of the genome-informed risk assessment | Baseline to 6 months post return of results to participant
  Number of new health care actions will be measured by electronic health record data and participant-reported outcomes through a REDCap survey. Pre-specified actions will include a condition-specific composite of new encounters, clinical orders, or specialty referrals for clinical evaluation associated with the condition(s), placed by a provider within 6 months of result disclosure.

SECONDARY OUTCOMES:
Number of newly diagnosed conditions after return of the genome-informed risk assessment | 6 months and 12 months post return of results to participant
  Number of newly diagnosed conditions included in the eMERGE study will be measured by data from participant electronic health records
Number of risk-reducing interventions after return of the genome-informed risk assessment | 6 months and 12 months post return of results to participant
  Number of risk-reducing interventions will be measured by REDCap survey along with data from participant electronic health records

CONTACTS AND LOCATIONS:
Overall Officials: Josh Peterson, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (12):
- United States (12):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Mountain Park Health Center, Tempe, Arizona
  - Northwestern, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roden DM, Pulley JM, Basford MA, Bernard GR, Clayton EW, Balser JR, Masys DR. Development of a large-scale de-identified DNA biobank to enable personalized medicine. Clin Pharmacol Ther. 2008 Sep;84(3):362-9. doi: 10.1038/clpt.2008.89. Epub 2008 May 21. PMID 18500243
- [Background] Pulley J, Clayton E, Bernard GR, Roden DM, Masys DR. Principles of human subjects protections applied in an opt-out, de-identified biobank. Clin Transl Sci. 2010 Feb;3(1):42-8. doi: 10.1111/j.1752-8062.2010.00175.x. PMID 20443953
- [Background] Bowton E, Field JR, Wang S, Schildcrout JS, Van Driest SL, Delaney JT, Cowan J, Weeke P, Mosley JD, Wells QS, Karnes JH, Shaffer C, Peterson JF, Denny JC, Roden DM, Pulley JM. Biobanks and electronic medical records: enabling cost-effective research. Sci Transl Med. 2014 Apr 30;6(234):234cm3. doi: 10.1126/scitranslmed.3008604. PMID 24786321
- [Background] Pulley JM, Brace MM, Bernard GR, Masys DR. Attitudes and perceptions of patients towards methods of establishing a DNA biobank. Cell Tissue Bank. 2008 Mar;9(1):55-65. doi: 10.1007/s10561-007-9051-2. Epub 2007 Oct 25. PMID 17960495
- [Background] Rosenbloom ST, Madison JL, Brothers KB, Bowton EA, Clayton EW, Malin BA, Roden DM, Pulley J. Ethical and practical challenges to studying patients who opt out of large-scale biorepository research. J Am Med Inform Assoc. 2013 Dec;20(e2):e221-5. doi: 10.1136/amiajnl-2013-001937. Epub 2013 Jul 25. PMID 23886923
- [Background] Bowton EA, Collier SP, Wang X, Sutcliffe CB, Van Driest SL, Couch LJ, Herrera M, Jerome RN, Slebos RJ, Alborn WE, Liebler DC, McNaughton CD, Mernaugh RL, Wells QS, Brown NJ, Roden DM, Pulley JM. Phenotype-Driven Plasma Biobanking Strategies and Methods. J Pers Med. 2015 May 14;5(2):140-52. doi: 10.3390/jpm5020140. PMID 26110578
- [Background] Brothers KB, Westbrook MJ, Wright MF, Myers JA, Morrison DR, Madison JL, Pulley JM, Clayton EW. Patient awareness and approval for an opt-out genomic biorepository. Per Med. 2013 Jun;10(4):10.2217/pme.13.34. doi: 10.2217/pme.13.34. PMID 24416062
- [Background] Pulley JM, Denny JC, Peterson JF, Bernard GR, Vnencak-Jones CL, Ramirez AH, Delaney JT, Bowton E, Brothers K, Johnson K, Crawford DC, Schildcrout J, Masys DR, Dilks HH, Wilke RA, Clayton EW, Shultz E, Laposata M, McPherson J, Jirjis JN, Roden DM. Operational implementation of prospective genotyping for personalized medicine: the design of the Vanderbilt PREDICT project. Clin Pharmacol Ther. 2012 Jul;92(1):87-95. doi: 10.1038/clpt.2011.371. Epub 2012 May 16. PMID 22588608
- [Background] Delaney JT, Ramirez AH, Bowton E, Pulley JM, Basford MA, Schildcrout JS, Shi Y, Zink R, Oetjens M, Xu H, Cleator JH, Jahangir E, Ritchie MD, Masys DR, Roden DM, Crawford DC, Denny JC. Predicting clopidogrel response using DNA samples linked to an electronic health record. Clin Pharmacol Ther. 2012 Feb;91(2):257-63. doi: 10.1038/clpt.2011.221. Epub 2011 Dec 21. PMID 22190063
- [Background] Karnes JH, Van Driest S, Bowton EA, Weeke PE, Mosley JD, Peterson JF, Denny JC, Roden DM. Using systems approaches to address challenges for clinical implementation of pharmacogenomics. Wiley Interdiscip Rev Syst Biol Med. 2014 Mar-Apr;6(2):125-35. doi: 10.1002/wsbm.1255. Epub 2013 Dec 6. PMID 24319008
- [Background] Peterson JF, Bowton E, Field JR, Beller M, Mitchell J, Schildcrout J, Gregg W, Johnson K, Jirjis JN, Roden DM, Pulley JM, Denny JC. Electronic health record design and implementation for pharmacogenomics: a local perspective. Genet Med. 2013 Oct;15(10):833-41. doi: 10.1038/gim.2013.109. Epub 2013 Sep 5. PMID 24009000
- [Background] Schildcrout JS, Denny JC, Bowton E, Gregg W, Pulley JM, Basford MA, Cowan JD, Xu H, Ramirez AH, Crawford DC, Ritchie MD, Peterson JF, Masys DR, Wilke RA, Roden DM. Optimizing drug outcomes through pharmacogenetics: a case for preemptive genotyping. Clin Pharmacol Ther. 2012 Aug;92(2):235-42. doi: 10.1038/clpt.2012.66. Epub 2012 Jun 27. PMID 22739144
- [Background] Van Driest SL, Shi Y, Bowton EA, Schildcrout JS, Peterson JF, Pulley J, Denny JC, Roden DM. Clinically actionable genotypes among 10,000 patients with preemptive pharmacogenomic testing. Clin Pharmacol Ther. 2014 Apr;95(4):423-31. doi: 10.1038/clpt.2013.229. Epub 2013 Nov 19. PMID 24253661
- [Background] Harris PA, Scott KW, Lebo L, Hassan N, Lightner C, Pulley J. ResearchMatch: a national registry to recruit volunteers for clinical research. Acad Med. 2012 Jan;87(1):66-73. doi: 10.1097/ACM.0b013e31823ab7d2. PMID 22104055
- [Background] Danciu I, Cowan JD, Basford M, Wang X, Saip A, Osgood S, Shirey-Rice J, Kirby J, Harris PA. Secondary use of clinical data: the Vanderbilt approach. J Biomed Inform. 2014 Dec;52:28-35. doi: 10.1016/j.jbi.2014.02.003. Epub 2014 Feb 14. PMID 24534443
- [Background] Rosenbloom ST, Harris P, Pulley J, Basford M, Grant J, DuBuisson A, Rothman RL. The Mid-South clinical Data Research Network. J Am Med Inform Assoc. 2014 Jul-Aug;21(4):627-32. doi: 10.1136/amiajnl-2014-002745. Epub 2014 May 12. PMID 24821742
- [Background] Byrne DW, Biaggioni I, Bernard GR, Helmer TT, Boone LR, Pulley JM, Edwards T, Dittus RS. Clinical and translational research studios: a multidisciplinary internal support program. Acad Med. 2012 Aug;87(8):1052-9. doi: 10.1097/ACM.0b013e31825d29d4. PMID 22722360
- [Background] Bernard GR, Harris PA, Pulley JM, Benjamin DK, Michael J, Ford DE, Hanley DF, Selker HP, Wilkins CH. A collaborative, academic approach to optimizing the national clinical research infrastructure: The first year of the Trial Innovation Network. J Clin Transl Sci. 2018 Aug;2(4):187-192. doi: 10.1017/cts.2018.319. Epub 2018 Nov 27. PMID 31011433
- [Background] Joosten YA, Israel TL, Williams NA, Boone LR, Schlundt DG, Mouton CP, Dittus RS, Bernard GR, Wilkins CH. Community Engagement Studios: A Structured Approach to Obtaining Meaningful Input From Stakeholders to Inform Research. Acad Med. 2015 Dec;90(12):1646-50. doi: 10.1097/ACM.0000000000000794. PMID 26107879
- [Background] Pulley JM, Harris PA, Yarbrough T, Swafford J, Edwards T, Bernard GR. An informatics-based tool to assist researchers in initiating research at an academic medical center: Vanderbilt Customized Action Plan. Acad Med. 2010 Jan;85(1):164-8. doi: 10.1097/ACM.0b013e3181c481bf. PMID 20042844
- [Background] Kirby JC, Speltz P, Rasmussen LV, Basford M, Gottesman O, Peissig PL, Pacheco JA, Tromp G, Pathak J, Carrell DS, Ellis SB, Lingren T, Thompson WK, Savova G, Haines J, Roden DM, Harris PA, Denny JC. PheKB: a catalog and workflow for creating electronic phenotype algorithms for transportability. J Am Med Inform Assoc. 2016 Nov;23(6):1046-1052. doi: 10.1093/jamia/ocv202. Epub 2016 Mar 28. PMID 27026615
- [Background] Mo H, Thompson WK, Rasmussen LV, Pacheco JA, Jiang G, Kiefer R, Zhu Q, Xu J, Montague E, Carrell DS, Lingren T, Mentch FD, Ni Y, Wehbe FH, Peissig PL, Tromp G, Larson EB, Chute CG, Pathak J, Denny JC, Speltz P, Kho AN, Jarvik GP, Bejan CA, Williams MS, Borthwick K, Kitchner TE, Roden DM, Harris PA. Desiderata for computable representations of electronic health records-driven phenotype algorithms. J Am Med Inform Assoc. 2015 Nov;22(6):1220-30. doi: 10.1093/jamia/ocv112. Epub 2015 Sep 5. PMID 26342218
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901
- [Background] Goldstein JI, Crenshaw A, Carey J, Grant GB, Maguire J, Fromer M, O'Dushlaine C, Moran JL, Chambert K, Stevens C; Swedish Schizophrenia Consortium; ARRA Autism Sequencing Consortium; Sklar P, Hultman CM, Purcell S, McCarroll SA, Sullivan PF, Daly MJ, Neale BM. zCall: a rare variant caller for array-based genotyping: genetics and population analysis. Bioinformatics. 2012 Oct 1;28(19):2543-5. doi: 10.1093/bioinformatics/bts479. Epub 2012 Jul 27. PMID 22843986
- [Background] Korn JM, Kuruvilla FG, McCarroll SA, Wysoker A, Nemesh J, Cawley S, Hubbell E, Veitch J, Collins PJ, Darvishi K, Lee C, Nizzari MM, Gabriel SB, Purcell S, Daly MJ, Altshuler D. Integrated genotype calling and association analysis of SNPs, common copy number polymorphisms and rare CNVs. Nat Genet. 2008 Oct;40(10):1253-60. doi: 10.1038/ng.237. Epub 2008 Sep 7. PMID 18776909
- [Background] Wilkins CH, Mapes BM, Jerome RN, Villalta-Gil V, Pulley JM, Harris PA. Understanding What Information Is Valued By Research Participants, And Why. Health Aff (Millwood). 2019 Mar;38(3):399-407. doi: 10.1377/hlthaff.2018.05046. PMID 30830824
- [Background] Khera AV, Chaffin M, Aragam KG, Haas ME, Roselli C, Choi SH, Natarajan P, Lander ES, Lubitz SA, Ellinor PT, Kathiresan S. Genome-wide polygenic scores for common diseases identify individuals with risk equivalent to monogenic mutations. Nat Genet. 2018 Sep;50(9):1219-1224. doi: 10.1038/s41588-018-0183-z. Epub 2018 Aug 13. PMID 30104762
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2019 Sep 10;74(10):1376-1414. doi: 10.1016/j.jacc.2019.03.009. Epub 2019 Mar 17. PMID 30894319
- [Background] Kanis JA, Johnell O, Oden A, Johansson H, McCloskey E. FRAX and the assessment of fracture probability in men and women from the UK. Osteoporos Int. 2008 Apr;19(4):385-97. doi: 10.1007/s00198-007-0543-5. Epub 2008 Feb 22. PMID 18292978
- [Background] Khera AV, Emdin CA, Drake I, Natarajan P, Bick AG, Cook NR, Chasman DI, Baber U, Mehran R, Rader DJ, Fuster V, Boerwinkle E, Melander O, Orho-Melander M, Ridker PM, Kathiresan S. Genetic Risk, Adherence to a Healthy Lifestyle, and Coronary Disease. N Engl J Med. 2016 Dec 15;375(24):2349-2358. doi: 10.1056/NEJMoa1605086. Epub 2016 Nov 13. PMID 27959714
- [Background] Mega JL, Stitziel NO, Smith JG, Chasman DI, Caulfield M, Devlin JJ, Nordio F, Hyde C, Cannon CP, Sacks F, Poulter N, Sever P, Ridker PM, Braunwald E, Melander O, Kathiresan S, Sabatine MS. Genetic risk, coronary heart disease events, and the clinical benefit of statin therapy: an analysis of primary and secondary prevention trials. Lancet. 2015 Jun 6;385(9984):2264-2271. doi: 10.1016/S0140-6736(14)61730-X. Epub 2015 Mar 4. PMID 25748612
- [Background] Mostafavi H, Harpak A, Agarwal I, Conley D, Pritchard JK, Przeworski M. Variable prediction accuracy of polygenic scores within an ancestry group. Elife. 2020 Jan 30;9:e48376. doi: 10.7554/eLife.48376. PMID 31999256
- [Background] Khera AV, Chaffin M, Zekavat SM, Collins RL, Roselli C, Natarajan P, Lichtman JH, D'Onofrio G, Mattera J, Dreyer R, Spertus JA, Taylor KD, Psaty BM, Rich SS, Post W, Gupta N, Gabriel S, Lander E, Ida Chen YD, Talkowski ME, Rotter JI, Krumholz HM, Kathiresan S. Whole-Genome Sequencing to Characterize Monogenic and Polygenic Contributions in Patients Hospitalized With Early-Onset Myocardial Infarction. Circulation. 2019 Mar 26;139(13):1593-1602. doi: 10.1161/CIRCULATIONAHA.118.035658. PMID 30586733
- [Background] Weigl K, Chang-Claude J, Knebel P, Hsu L, Hoffmeister M, Brenner H. Strongly enhanced colorectal cancer risk stratification by combining family history and genetic risk score. Clin Epidemiol. 2018 Jan 19;10:143-152. doi: 10.2147/CLEP.S145636. eCollection 2018. PMID 29403313
- [Background] Murray MF, Giovanni MA, Klinger E, George E, Marinacci L, Getty G, Brawarsky P, Rocha B, Orav EJ, Bates DW, Haas JS. Comparing electronic health record portals to obtain patient-entered family health history in primary care. J Gen Intern Med. 2013 Dec;28(12):1558-64. doi: 10.1007/s11606-013-2442-0. Epub 2013 Apr 16. PMID 23588670
- [Background] Guttmacher AE, Collins FS, Carmona RH. The family history--more important than ever. N Engl J Med. 2004 Nov 25;351(22):2333-6. doi: 10.1056/NEJMsb042979. No abstract available. PMID 15564550
- [Background] Krist AH, Beasley JW, Crosson JC, Kibbe DC, Klinkman MS, Lehmann CU, Fox CH, Mitchell JM, Mold JW, Pace WD, Peterson KA, Phillips RL, Post R, Puro J, Raddock M, Simkus R, Waldren SE. Electronic health record functionality needed to better support primary care. J Am Med Inform Assoc. 2014 Sep-Oct;21(5):764-71. doi: 10.1136/amiajnl-2013-002229. Epub 2014 Jan 15. PMID 24431335
- [Background] Hulse NC, Ranade-Kharkar P, Post H, Wood GM, Williams MS, Haug PJ. Development and early usage patterns of a consumer-facing family health history tool. AMIA Annu Symp Proc. 2011;2011:578-87. Epub 2011 Oct 22. PMID 22195113
- [Background] Denny JC, Crawford DC, Ritchie MD, Bielinski SJ, Basford MA, Bradford Y, Chai HS, Bastarache L, Zuvich R, Peissig P, Carrell D, Ramirez AH, Pathak J, Wilke RA, Rasmussen L, Wang X, Pacheco JA, Kho AN, Hayes MG, Weston N, Matsumoto M, Kopp PA, Newton KM, Jarvik GP, Li R, Manolio TA, Kullo IJ, Chute CG, Chisholm RL, Larson EB, McCarty CA, Masys DR, Roden DM, de Andrade M. Variants near FOXE1 are associated with hypothyroidism and other thyroid conditions: using electronic medical records for genome- and phenome-wide studies. Am J Hum Genet. 2011 Oct 7;89(4):529-42. doi: 10.1016/j.ajhg.2011.09.008. PMID 21981779
- [Background] Denny JC, Ritchie MD, Basford MA, Pulley JM, Bastarache L, Brown-Gentry K, Wang D, Masys DR, Roden DM, Crawford DC. PheWAS: demonstrating the feasibility of a phenome-wide scan to discover gene-disease associations. Bioinformatics. 2010 May 1;26(9):1205-10. doi: 10.1093/bioinformatics/btq126. Epub 2010 Mar 24. PMID 20335276
- [Background] Denny JC, Bastarache L, Ritchie MD, Carroll RJ, Zink R, Mosley JD, Field JR, Pulley JM, Ramirez AH, Bowton E, Basford MA, Carrell DS, Peissig PL, Kho AN, Pacheco JA, Rasmussen LV, Crosslin DR, Crane PK, Pathak J, Bielinski SJ, Pendergrass SA, Xu H, Hindorff LA, Li R, Manolio TA, Chute CG, Chisholm RL, Larson EB, Jarvik GP, Brilliant MH, McCarty CA, Kullo IJ, Haines JL, Crawford DC, Masys DR, Roden DM. Systematic comparison of phenome-wide association study of electronic medical record data and genome-wide association study data. Nat Biotechnol. 2013 Dec;31(12):1102-10. doi: 10.1038/nbt.2749. PMID 24270849
- [Background] Ritchie MD, Denny JC, Zuvich RL, Crawford DC, Schildcrout JS, Bastarache L, Ramirez AH, Mosley JD, Pulley JM, Basford MA, Bradford Y, Rasmussen LV, Pathak J, Chute CG, Kullo IJ, McCarty CA, Chisholm RL, Kho AN, Carlson CS, Larson EB, Jarvik GP, Sotoodehnia N; Cohorts for Heart and Aging Research in Genomic Epidemiology (CHARGE) QRS Group; Manolio TA, Li R, Masys DR, Haines JL, Roden DM. Genome- and phenome-wide analyses of cardiac conduction identifies markers of arrhythmia risk. Circulation. 2013 Apr 2;127(13):1377-85. doi: 10.1161/CIRCULATIONAHA.112.000604. Epub 2013 Mar 5. PMID 23463857
- [Background] Simonti CN, Vernot B, Bastarache L, Bottinger E, Carrell DS, Chisholm RL, Crosslin DR, Hebbring SJ, Jarvik GP, Kullo IJ, Li R, Pathak J, Ritchie MD, Roden DM, Verma SS, Tromp G, Prato JD, Bush WS, Akey JM, Denny JC, Capra JA. The phenotypic legacy of admixture between modern humans and Neandertals. Science. 2016 Feb 12;351(6274):737-41. doi: 10.1126/science.aad2149. PMID 26912863
- [Background] Rasmussen-Torvik LJ, Stallings SC, Gordon AS, Almoguera B, Basford MA, Bielinski SJ, Brautbar A, Brilliant MH, Carrell DS, Connolly JJ, Crosslin DR, Doheny KF, Gallego CJ, Gottesman O, Kim DS, Leppig KA, Li R, Lin S, Manzi S, Mejia AR, Pacheco JA, Pan V, Pathak J, Perry CL, Peterson JF, Prows CA, Ralston J, Rasmussen LV, Ritchie MD, Sadhasivam S, Scott SA, Smith M, Vega A, Vinks AA, Volpi S, Wolf WA, Bottinger E, Chisholm RL, Chute CG, Haines JL, Harley JB, Keating B, Holm IA, Kullo IJ, Jarvik GP, Larson EB, Manolio T, McCarty CA, Nickerson DA, Scherer SE, Williams MS, Roden DM, Denny JC. Design and anticipated outcomes of the eMERGE-PGx project: a multicenter pilot for preemptive pharmacogenomics in electronic health record systems. Clin Pharmacol Ther. 2014 Oct;96(4):482-9. doi: 10.1038/clpt.2014.137. Epub 2014 Jun 24. PMID 24960519
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Wu RR, Himmel TL, Buchanan AH, Powell KP, Hauser ER, Ginsburg GS, Henrich VC, Orlando LA. Quality of family history collection with use of a patient facing family history assessment tool. BMC Fam Pract. 2014 Feb 13;15:31. doi: 10.1186/1471-2296-15-31. PMID 24520818
- [Background] Beadles CA, Ryanne Wu R, Himmel T, Buchanan AH, Powell KP, Hauser E, Henrich VC, Ginsburg GS, Orlando LA. Providing patient education: impact on quantity and quality of family health history collection. Fam Cancer. 2014 Jun;13(2):325-32. doi: 10.1007/s10689-014-9701-z. PMID 24515581
- [Background] Wu RR, Orlando LA, Himmel TL, Buchanan AH, Powell KP, Hauser ER, Agbaje AB, Henrich VC, Ginsburg GS. Patient and primary care provider experience using a family health history collection, risk stratification, and clinical decision support tool: a type 2 hybrid controlled implementation-effectiveness trial. BMC Fam Pract. 2013 Aug 6;14:111. doi: 10.1186/1471-2296-14-111. PMID 23915256
- [Background] O'Neill SM, Rubinstein WS, Wang C, Yoon PW, Acheson LS, Rothrock N, Starzyk EJ, Beaumont JL, Galliher JM, Ruffin MT 4th; Family Healthware Impact Trial group. Familial risk for common diseases in primary care: the Family Healthware Impact Trial. Am J Prev Med. 2009 Jun;36(6):506-14. doi: 10.1016/j.amepre.2009.03.002. PMID 19460658
- [Background] Hripcsak G, Shang N, Peissig PL, Rasmussen LV, Liu C, Benoit B, Carroll RJ, Carrell DS, Denny JC, Dikilitas O, Gainer VS, Howell KM, Klann JG, Kullo IJ, Lingren T, Mentch FD, Murphy SN, Natarajan K, Pacheco JA, Wei WQ, Wiley K, Weng C. Facilitating phenotype transfer using a common data model. J Biomed Inform. 2019 Aug;96:103253. doi: 10.1016/j.jbi.2019.103253. Epub 2019 Jul 17. PMID 31325501
- [Background] Nguyen XT, Quaden RM, Song RJ, Ho YL, Honerlaw J, Whitbourne S, DuVall SL, Deen J, Pyarajan S, Moser J, Huang GD, Muralidhar S, Concato J, Tsao PS, O'Donnell CJ, Wilson PWF, Djousse L, Gagnon DR, Gaziano JM, Cho K. Baseline Characterization and Annual Trends of Body Mass Index for a Mega-Biobank Cohort of US Veterans 2011-2017. J Health Res Rev Dev Ctries. 2018;5(2):98-107. PMID 33117892
- [Background] Li M, Scaiano M, El Emam K, Malin BA. Efficient Active Learning for Electronic Medical Record De-identification. AMIA Jt Summits Transl Sci Proc. 2019 May 6;2019:462-471. eCollection 2019. PMID 31259000
- [Background] Liu Y, Wan Z, Xia W, Kantarcioglu M, Vorobeychik Y, Clayton EW, Kho A, Carrell D, Malin BA. Detecting the Presence of an Individual in Phenotypic Summary Data. AMIA Annu Symp Proc. 2018 Dec 5;2018:760-769. eCollection 2018. PMID 30815118
- [Background] Xia W, Wan Z, Yin Z, Gaupp J, Liu Y, Clayton EW, Kantarcioglu M, Vorobeychik Y, Malin BA. It's all in the timing: calibrating temporal penalties for biomedical data sharing. J Am Med Inform Assoc. 2018 Jan 1;25(1):25-31. doi: 10.1093/jamia/ocx101. PMID 29036325
- [Background] Prasser F, Gaupp J, Wan Z, Xia W, Vorobeychik Y, Kantarcioglu M, Kuhn K, Malin B. An Open Source Tool for Game Theoretic Health Data De-Identification. AMIA Annu Symp Proc. 2018 Apr 16;2017:1430-1439. eCollection 2017. PMID 29854212
- [Background] Heatherly R, Rasmussen LV, Peissig PL, Pacheco JA, Harris P, Denny JC, Malin BA. A multi-institution evaluation of clinical profile anonymization. J Am Med Inform Assoc. 2016 Apr;23(e1):e131-7. doi: 10.1093/jamia/ocv154. Epub 2015 Nov 13. PMID 26567325
- [Background] El Emam K, Rodgers S, Malin B. Anonymising and sharing individual patient data. BMJ. 2015 Mar 20;350:h1139. doi: 10.1136/bmj.h1139. PMID 25794882
- [Background] Xia W, Heatherly R, Ding X, Li J, Malin BA. R-U policy frontiers for health data de-identification. J Am Med Inform Assoc. 2015 Sep;22(5):1029-41. doi: 10.1093/jamia/ocv004. Epub 2015 Apr 24. PMID 25911674
- [Background] Wan Z, Vorobeychik Y, Xia W, Clayton EW, Kantarcioglu M, Ganta R, Heatherly R, Malin BA. A game theoretic framework for analyzing re-identification risk. PLoS One. 2015 Mar 25;10(3):e0120592. doi: 10.1371/journal.pone.0120592. eCollection 2015. PMID 25807380
- [Background] Loh PR, Danecek P, Palamara PF, Fuchsberger C, A Reshef Y, K Finucane H, Schoenherr S, Forer L, McCarthy S, Abecasis GR, Durbin R, L Price A. Reference-based phasing using the Haplotype Reference Consortium panel. Nat Genet. 2016 Nov;48(11):1443-1448. doi: 10.1038/ng.3679. Epub 2016 Oct 3. PMID 27694958
- [Background] Campion TR Jr, Sholle ET, Davila MA Jr. Generalizable Middleware to Support Use of REDCap Dynamic Data Pull for Integrating Clinical and Research Data. AMIA Jt Summits Transl Sci Proc. 2017 Jul 26;2017:76-81. eCollection 2017. PMID 28815111
- [Background] Sperber NR, Carpenter JS, Cavallari LH, J Damschroder L, Cooper-DeHoff RM, Denny JC, Ginsburg GS, Guan Y, Horowitz CR, Levy KD, Levy MA, Madden EB, Matheny ME, Pollin TI, Pratt VM, Rosenman M, Voils CI, W Weitzel K, Wilke RA, Ryanne Wu R, Orlando LA. Challenges and strategies for implementing genomic services in diverse settings: experiences from the Implementing GeNomics In pracTicE (IGNITE) network. BMC Med Genomics. 2017 May 22;10(1):35. doi: 10.1186/s12920-017-0273-2. PMID 28532511
- [Derived] Connolly JJ, Berner ES, Smith M, Levy S, Terek S, Harr M, Karavite D, Suckiel S, Holm IA, Dufendach K, Nelson C, Khan A, Chisholm RL, Allworth A, Wei WQ, Bland HT, Clayton EW, Soper ER, Linder JE, Limdi NA, Miller A, Nigbur S, Bangash H, Hamed M, Sherafati A, Lewis ACF, Perez E, Orlando LA, Rakhra-Burris TK, Al-Dulaimi M, Cifric S, Scherr CL, Wynn J, Hakonarson H, Sabatello M. Education and electronic medical records and genomics network, challenges, and lessons learned from a large-scale clinical trial using polygenic risk scores. Genet Med. 2023 Sep;25(9):100906. doi: 10.1016/j.gim.2023.100906. Epub 2023 May 26. PMID 37246632
- [Derived] Linder JE, Allworth A, Bland HT, Caraballo PJ, Chisholm RL, Clayton EW, Crosslin DR, Dikilitas O, DiVietro A, Esplin ED, Forman S, Freimuth RR, Gordon AS, Green R, Harden MV, Holm IA, Jarvik GP, Karlson EW, Labrecque S, Lennon NJ, Limdi NA, Mittendorf KF, Murphy SN, Orlando L, Prows CA, Rasmussen LV, Rasmussen-Torvik L, Rowley R, Sawicki KT, Schmidlen T, Terek S, Veenstra D, Velez Edwards DR, Absher D, Abul-Husn NS, Alsip J, Bangash H, Beasley M, Below JE, Berner ES, Booth J, Chung WK, Cimino JJ, Connolly J, Davis P, Devine B, Fullerton SM, Guiducci C, Habrat ML, Hain H, Hakonarson H, Harr M, Haverfield E, Hernandez V, Hoell C, Horike-Pyne M, Hripcsak G, Irvin MR, Kachulis C, Karavite D, Kenny EE, Khan A, Kiryluk K, Korf B, Kottyan L, Kullo IJ, Larkin K, Liu C, Malolepsza E, Manolio TA, May T, McNally EM, Mentch F, Miller A, Mooney SD, Murali P, Mutai B, Muthu N, Namjou B, Perez EF, Puckelwartz MJ, Rakhra-Burris T, Roden DM, Rosenthal EA, Saadatagah S, Sabatello M, Schaid DJ, Schultz B, Seabolt L, Shaibi GQ, Sharp RR, Shirts B, Smith ME, Smoller JW, Sterling R, Suckiel SA, Thayer J, Tiwari HK, Trinidad SB, Walunas T, Wei WQ, Wells QS, Weng C, Wiesner GL, Wiley K; eMERGE Consortium; Peterson JF. Returning integrated genomic risk and clinical recommendations: The eMERGE study. Genet Med. 2023 Apr;25(4):100006. doi: 10.1016/j.gim.2023.100006. Epub 2023 Jan 6. PMID 36621880